CLINICAL TRIAL: NCT03654560
Title: Efficacy and Safety of HemoStyp as an Adjunct for Management of Secondary Hemostasis in the Operative Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United Health Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UHP001
Record Dates: First submitted 2018-08-27; First posted 2018-08-31 (Actual); Results first posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2019-10

CONDITIONS: Hemostasis; Bleeding
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- HemoStyp (Active Comparator): Subjects with an appropriate target bleeding site will have Hemostyp applied in accordance to instructions for use.
  Interventions: Device: HemoStyp
- Surgicel (Active Comparator): Subjects with an appropriate target bleeding site will have Surgicel applied in accordance to instructions for use.
  Interventions: Device: Surgicel

INTERVENTIONS:
Device: HemoStyp — During elective surgical procedure (non-laparoscopic thoracic, cardiac, abdominal, or vascular surgery) subject has mild to moderate soft tissue, vascular or parenchymal bleeding present at target bleeding site after primary standard conventional surgical hemostatic methods are proven to be ineffective or impractical will have Hemostyp applied in accordance to instructions for use.
  Arms: HemoStyp
Device: Surgicel — During elective surgical procedure (non-laparoscopic thoracic, cardiac, abdominal, or vascular surgery) subject has mild to moderate soft tissue, vascular or parenchymal bleeding present at target bleeding site after primary standard conventional surgical hemostatic methods are proven to be ineffective or impractical will have Surgicel applied in accordance to instructions for use.
  Arms: Surgicel

SUMMARY:
The purpose of the study is to assess efficacy and safety of HemoStyp as an adjunct for management of secondary hemostasis in the operative setting.

DETAILED DESCRIPTION:
This study is a prospective, non-inferiority, multi-center, randomized, open-label trial to compare HemoStyp with Surgicel® in the management of bleeding during surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Elective procedure (non-laparoscopic thoracic, cardiac, abdominal, or vascular surgery);
2. At time of surgery has mild to moderate soft tissue, vascular or parenchymal bleeding present at target bleeding site after primary standard conventional surgical hemostatic methods are proven to be ineffective or impractical;
3. Ages: Pediatric subjects 2 years to 17 years of age and adult subjects 18 years of age or older; and
4. Subjects or parent or legal guardian of the subject who are willing and able to sign consent.

Exclusion Criteria:

1. Physical or psychological condition which would impair study participation;
2. Indications for emergency surgery;
3. Pre-operative laboratory findings of a hematologic disorder;
4. Subjects with history of moderate to severe allergies;
5. Subjects undergoing minimally invasive laparoscopic surgery;
6. Subjects who will require platelet or fresh frozen plasma transfusion during surgery;
7. Subjects who are pregnant or breast-feeding at the time of surgery; or
8. Subjects on P2Y12 platelet inhibitor (Plavix) less than 5 days prior to surgery, warfarin or Xa inhibitors not withheld per standard protocols for the management of anticoagulants pre-operatively.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2018-12-28 (Actual); Primary Completion 2019-08-05 (Actual); Study Completion 2019-09-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Raymond Schaerf, Burbank, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HemoStyp | Surgicel
Started | 118 | 118
Completed | 114 | 117
Not Completed | 4 | 1
Not completed — Death | 3 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HemoStyp | Surgicel | Total
Number analyzed (Participants) | 118 | 118 | 236
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.89 (16.13) | 61.48 (16.48) | 60.19 (16.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 45 | 97
  Male | 66 | 73 | 139
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 26 | 57
  Not Hispanic or Latino | 87 | 92 | 179
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 10 | 6 | 16
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 5 | 3 | 8
  White | 74 | 86 | 160
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 28 | 22 | 50
Height [Mean (Standard Deviation); unit: cm] | 164.84 (19.59) | 168.55 (15.5) | 166.69 (19.59)
Weight [Mean (Standard Deviation); unit: kg] | 79.94 (38.62) | 86.48 (49.88) | 83.24 (38.62)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 124.11 (25.14) | 124.53 (26.75) | 124.26 (26.36)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 67.34 (16.87) | 67.48 (16.09) | 67.45 (16.87)
Heart Rate [Mean (Standard Deviation); unit: Beats Per minute] | 71.26 (13.87) | 71.89 (13.12) | 71.54 (13.67)
Hemoglobin [Mean (Standard Deviation); unit: grams per deciliter] | 12.37 (2.83) | 12.14 (2.69) | 12.25 (2.83)
Hematocrit [Mean (Standard Deviation); unit: percentage] | 40.18 (26.52) | 36.16 (7.71) | 38.15 (26.52)
Platelet Count [Mean (Standard Deviation); unit: platelets per micro liter of blood] | 212.83 (92.5) | 221.81 (99.45) | 217.36 (92.5)
Type of Surgery [Count of Participants; unit: Participants]
  Abdominal Surgery | 35 | 37 | 72
  Thoracic Surgery | 32 | 38 | 70
  Vascular Surgery | 51 | 43 | 94
Lewis Bleeding Scale Grade [Count of Participants; unit: Participants] — Investigator rated the intensity of the bleeding at the target bleeding site (TBS) according to the validated bleeding scale (Lewis 2017) shown below.
  Lewis Bleeding Scale Description:
  Grade 1 is an ooze or intermittent flow with capillary-like bleeding, described as mild bleeding with >1.0-5.0 milliliters per minutes (ML/Min) blood loss.
  Grade 2 is a continuous flow, venule and arteriolar-like bleeding described as moderate bleeding with >5.0-10.0 ML/Min blood loss
  Participants
    Lewis Bleeding Scale Grade 1 | 61 | 73 | 134
    Lewis Bleeding Scale Grade 2 | 57 | 45 | 102

OUTCOME MEASURES:

1. Primary Outcome: The Time to Hemostasis Measured From Start of Study Treatment to the Achievement of Hemostasis at the Target Bleeding Site (TBS), or to the End of the 10-minute Observation Period.
Description: The time to hemostasis was measured from start of study treatment to the achievement of hemostasis at the target bleeding site (TBS), or to the end of the 10-minute observation period. The time to hemostasis was considered as censored at the end of the 10-minute observation period. Time to hemostasis was quantified in minutes according to its nominal time point. When re-bleeding occurred, and the cessation of bleeding is again achieved at a later time point, the effective time to hemostasis was the latter time point. The time to hemostasis was the time from start of study treatment to that last effective hemostatic time point.
Time Frame: 10 minutes
Measure: Median (95% Confidence Interval); unit: seconds
Arm/Group | HemoStyp | Surgicel
Number analyzed (Participants) | 118 | 118
seconds | 36 [31 to 47] | 67 [57 to 89]

2. Secondary Outcome: Percentage of Subjects Achieving Hemostasis Between 2 Minutes and 10 Minutes
Description: Percentage of subjects achieving hemostasis at the target bleeding site at 2 minutes, 5 minutes and 10 minutes following the start of study treatment.
Time Frame: Between 2 minutes and 10 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | HemoStyp | Surgicel
Number analyzed (Participants) | 118 | 118
Participants
  2 minutes | 118 | 96
  5 minutes | 118 | 110
  10 minutes | 118 | 112

3. Secondary Outcome: Rate of Subjects Achieving Intraoperative Hemostasis at the Target Bleeding Site
Description: Percentage of subjects with intraoperative hemostasis at the target bleeding site during the intraoperative period. The intraoperative period started when the first cut was made to the patient and ended when the operative field was closed and dressed.
Time Frame: Intraoperative period
Measure: Count of Participants; unit: Participants
Arm/Group | HemoStyp | Surgicel
Number analyzed (Participants) | 118 | 118
Participants | 118 | 112

4. Secondary Outcome: Rate of Subjects With Intraoperative Re-bleeding From the Target Bleeding Site
Description: Percentage of subjects with intraoperative re-bleeding from the target bleeding site post hemostasis
Time Frame: Intraoperative period post hemostasis
Population: 6 subjects in the Surgicel cohort could not be analyzed because hemostasis was never obtained at the target bleeding site.
Measure: Count of Participants; unit: Participants
Arm/Group | HemoStyp | Surgicel
Number analyzed (Participants) | 118 | 112
Participants | 0 | 0

5. Secondary Outcome: Rate of Subjects Requiring Surgical Re-exploration up to 30 Days After Surgery for Re-bleeding From the Target Bleeding Site
Description: Postoperative re-bleeding from the target bleeding site requiring surgical re exploration up to 30 days after surgery.
Time Frame: 30 days
Population: 3 subjects in the HemoStyp cohort and 6 subjects in the Surgicel cohort did not finish the 30 day follow up so they were not included in the analysis population.
Measure: Count of Participants; unit: Participants
Arm/Group | HemoStyp | Surgicel
Number analyzed (Participants) | 115 | 112
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From treatment to 30 days.
Arm/Group | HemoStyp | Surgicel
All-Cause Mortality (participants affected / at risk) | 3/118 | 1/118
Serious Adverse Events (participants affected / at risk) | 1/118 | 0/118
Other Adverse Events (participants affected / at risk) | 0/118 | 4/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HemoStyp (N=118) | Surgicel (N=118)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Patient had pneumonia requiring hospitalization, not related to the study treatment.
Soft Tissue infection (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Necrotizing soft tissue infection at site of surgery, requiring abdominal wall debridement. Not related to the study treatment.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HemoStyp (N=118) | Surgicel (N=118)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) — Abdominal pain that resolved. Not related to the study treatment.
Pelvic Pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) — Pelvic Pain resolved, not related to the study treatment.
Bleeding Anterior Venous Fistula (Vascular disorders) | 0 (0) | 1 (1) — Bleeding of anterior venous fistula, not in the area of the treatment and not related to the study device.
Seroma (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Seroma not related to the study treatment.
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) — Constipation not related to the study treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-02): https://cdn.clinicaltrials.gov/large-docs/60/NCT03654560/Prot_SAP_000.pdf